CLINICAL TRIAL: NCT05805124
Title: Do Anesthesiologists Follow Belgian KCE Guidelines for Preoperative Evaluation in Patients Undergoing Non-emergency Surgery ?
Brief Title: Do Anesthesiologists Follow Belgian KCE Guidelines for Preoperative Evaluation?
Status: Completed | Type: Observational
Sponsor: Erasme University Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: SRB2023061
Record Dates: First submitted 2023-03-28; First posted 2023-04-07 (Actual); Last update posted 2023-08-30 (Actual); Status verified 2023-03

CONDITIONS: Surgery

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Diagnostic Test: Preop evaluation — All preop evaluations prescribed in the preadmission clinic will be recorded, especially:
  * renal function tests
  * hematologic tests
  * coagulation tests
  * hepatic function tests
  * ECG
  * cardiac function tests
  * pulmonary function tests
  * endocrine function tests

SUMMARY:
For more than 50 years it has been shown that preoperative evaluations by anesthesiologists include too many unnecessary tests. Many of the tests ordered do not change the management of the patients. One example are preoperative coagulation tests which rarely give relevant information and can be omitted if the patients have a negative structured bleeding questionnaire. This situation has lead to the publication of many guidelines on preoperative evaluation, one of the most comprehensive being the 2022 guidelines by the European Society of Cardiology for the preoperative evaluation of cardiac patients undergoing non-cardiac surgery.

In Belgium, an independent center of experts, the Kenniscentrum - Centre d'Expertise (KCE) was created to give expert and independent opinions on healthcare related subjects. These recommendations are often used by Belgian authorities to guide public health law and determine which medical procedures or tests are covered by the social security.

The KCE has published an extensive guide on preoperative evaluation of patients undergoing non-cardiac surgery (KCE Reports 280Bs. D/2016/10.273/102.) These guidelines are freely available, either in print version, on the dedicated Website or as an App, and have been extensively spread in the anesthesiology community. Laboratory tests not recommended in these guidelines are not covered by the social security if no solid reason is given in the medical chart.

In this retrospective study, adherence to the KCE guidelines on preoperative evaluations will be evaluated in a tertiary University hospital. All patients, scheduled for elective surgery, will be included for a period of 3 month. For every patient the recommended tests will be determined and compared to the actual tests prescribed by the anesthesiologist during the preadmission visit.

ELIGIBILITY:
Inclusion Criteria:

* All patients examined at the anesthesiology preadmission clinic during Oct 1st 2022 and december 31st 2022 and scheduled for elective surgery at Erasme University hospital under general or locoregional anesthesia

Exclusion Criteria:

* Non elective surgery
* Age < 18 years
* surgery under local anesthesia

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All patients scheduled for elective surgery under general or locoregional anesthesia at Erasme University hospital seen at the anesthesiology preadmission clinic during Oct 1st 2022 and Dec 31st 2022
Sampling Method: Non-Probability Sample
Enrollment: 2521 (Actual)
Dates: Start 2023-08-01 (Actual); Primary Completion 2023-08-25 (Actual); Study Completion 2023-08-29 (Actual)

PRIMARY OUTCOMES:
Adherence to KCE recommendations in percentage | 24 hours
  Every tests prescribed in the anesthesiology preadmission clinic will be compared to the KCE recommendations. Each test will be classified as "appropriate" or "not recommended". The percentage of adherence to the KCE guidelines will be reported for each test.

CONTACTS AND LOCATIONS:
Locations (1):
- Hôpital Universitaire de Bruxelles - Hôpital erasme, Brussels, Belgium

IPD SHARING:
Plan to Share IPD: No